CLINICAL TRIAL: NCT05966909
Title: Asymptomatic PICC-related Thrombosis in Cancer Patients: a Prospective Cohort Study of an Ultrasound-guided Approach.
Brief Title: Incidence and Clinical Progression of Asymptomatic PICC-Related Thrombosis in Solid Cancer Patients
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Principal Investigator, Luca Giuseppe Dalle Carbonare, Associate Professor, Azienda Ospedaliera Universitaria Integrata Verona
Other Study IDs: THROMBPICC
Record Dates: First submitted 2023-07-21; First posted 2023-08-01 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-08

CONDITIONS: Catheter Related Complication
Keywords: Catheter-related thrombosis; Peripherally inserted central catheter-ports; Cancer associated thrombosis; Upper extremities vein thrombosis
MeSH Terms: interventions — Ultrasonography, Doppler

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Solid cancer patients: Patients with solid cancer who underwent the placement of a PICC or PICC-PORT for chemotherapy.
  Interventions: Diagnostic Test: Doppler Ultrasound

INTERVENTIONS:
Diagnostic Test: Doppler Ultrasound — Ultrasound diagnosi of asymptomatic and symptomatic upper extremities vein thrombosis

SUMMARY:
In this prospective cohort study, the investigators evaluated the incidence of superficial vein thrombosis, deep vein thrombosis, and fibroblastic sleeve formation in solid cancer patients undergoing chemotherapy. The study aimed to shed light on the clinical progression of venous thrombosis in cancer patients with central venous catheters, with a particular focus on certain cancer types associated with a higher risk of venous thromboembolism (VTE).

The investigators believe that such findings hold significant clinical relevance as a substantial portion of the study population was affected by pancreatic cancer, a cancer type known to carry a high risk of thrombotic events. This research adds valuable insights into understanding asymptomatic PICC-related thrombosis in this specific subgroup of cancer patients, which can aid in developing effective management strategies for venous access in this challenging population.

The study employed an ultrasound-guided approach for follow-up at 30 and 90 days after catheter insertion, enabling us to detect and treat asymptomatic PICC-VTE in a timely manner. Identifying independent risk factors for catheter-related thrombosis, including age and cancer type, has further enhanced the clinical applicability of our findings.

DETAILED DESCRIPTION:
Managing venous access in cancer patients is challenging, and peripherally inserted central catheter-ports (PICC-ports) have emerged as a promising option for safety and efficacy. However, understanding the clinical progression of venous thrombosis in cancer patients with central venous catheters remains limited, especially in certain cancer types associated with a higher risk of venous thromboembolism (VTE).

In this prospective cohort study of solid cancer patients receiving chemotherapy, the investigators will evaluate the incidence of superficial vein thrombosis, deep vein thrombosis, and fibroblastic sleeve formation through ultrasound follow-up at 30 and 90 days after catheter insertion. The investigators will analyze clinical factors associated with PICC-related VTE (PICC-VTE) and compare incidence rates between PICC-ports and traditional PICCs.

Ultrasound follow-up is valuable for detecting asymptomatic PICC-VTE, enabling timely and effective initiation of therapy, especially in elderly patients and those with high-risk thrombotic cancers.

ELIGIBILITY:
Inclusion Criteria:

* patients with:

  1. a documented active malignancy;
  2. PICC or PORT placement for systemic chemotherapy;

Exclusion Criteria:

* patients with:

  1. a communication disorder;
  2. contraindications to anticoagulation therapy;
  3. hematopathy;
  4. expected survival of less than one month;
  5. were lost to follow-up.

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with solid cancer undergoing chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Catheter related thrombosis | 1 month and 3 months from baseline
  Symptomatic and asymptomatic upper extremities thrombosis

SECONDARY OUTCOMES:
PICC vs PICC-PORT | 1 month and 3 months from baseline
  Risk factors associated with Catheter related Thrombosis

CONTACTS AND LOCATIONS:
Overall Officials: Mattia Cominacini, MD, Study Director — Azienda Ospedaliera Universitaria Integrata Verona
Locations (1):
- Azienda Ospedaliera Universitaria Integrata, Verona, Italy

IPD SHARING:
Plan to Share IPD: No